CLINICAL TRIAL: NCT00584480
Title: Pilot Study of the Effect of Hyperbaric Oxygen Treatment on Behavioral and Biomarker Measures in Children With Autism
Acronym: HBOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200715202-1
Record Dates: First submitted 2007-12-22; First posted 2008-01-02 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Active Hyperbaric Oxygen Treatment (HBOT)
  Interventions: Other: Hyperbaric Oxygen Treatment (HBOT)

INTERVENTIONS:
Other: Hyperbaric Oxygen Treatment (HBOT) — 1.5 ATA at 100% Oxygen of HBOT

SUMMARY:
The purpose of this study is to increase the understanding of the effect of Hyperbaric Oxygen Treatment (HBOT) on the behavior and functioning of children with autism. The main goal of this study is to demonstrate that HBOT is safe and tolerable in autistic children, and to measure the effect of HBOT on specific chemicals in their blood that may play a role in the child's behavior.

DETAILED DESCRIPTION:
During the study's 20-week duration, all children will receive Hyperbaric Oxygen Treatment (HBOT) for two eight-week sessions, with a four week session between. Therefore, all children will participate in the study for 20 weeks, and will receive HBOT for 16 weeks. This is an open label study. This means that there will not be a placebo group in the study. All study participants will receive the same treatment of HBOT in a hard shell chamber. Normal air contains about 24% oxygen at a pressure of about 1 atmosphere absolute (ATA). The chamber will contain 100 percent oxygen at a pressure of 1.5 ATA, which is equivalent to the pressure at a depth of 15 feet in sea water. Each subject will complete the first 40 treatments during one hour sessions on 5 separate days in each of the first 8 weeks. They will then take a 4-week break before they begin their next 40 treatments, which will also occur during one hour sessions on 5 separate days in each of the last 8 weeks. The entire study will last 20 weeks. The child's behavior will be measured and evaluated at the MIND Institute at the beginning of the study, at week 8, and at week 20.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of DSM-IV defined autism and meets cut off for autism on the Autism Diagnostic Inventory-Revised (ADI-R) or Social Communication Questionnaire (SCQ) and the Autism Diagnostic Observation Scale (ADOS).
2. Age 3 to 8 years.
3. Nonverbal IQ of 50 or above.
4. Parental agreement to continue present dietary, behavioral or psychotropic drug treatment but not change treatment during 20 week intervention.

Exclusion Criteria:

1. Clinical evidence of seizure disorder
2. Active infection with fever
3. Fragile X or other known genetic cause of autism
4. Perinatal brain injury (e.g. cerebral palsy)
5. Previous adequate trial (at least 20 session) of HBOT
6. Inability to clear ears in the HBOT chambers

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Hendren, DO, Principal Investigator — University of California, Davis - M.I.N.D. Institute

REFERENCES:
- [Derived] Bent S, Bertoglio K, Ashwood P, Nemeth E, Hendren RL. Brief report: Hyperbaric oxygen therapy (HBOT) in children with autism spectrum disorder: a clinical trial. J Autism Dev Disord. 2012 Jun;42(6):1127-32. doi: 10.1007/s10803-011-1337-3. PMID 21818676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place between October 1, 2007 to April 24, 2009. Children between the ages of 3 and 8 with a diagnosis of Autism Spectrum Disorders (ASD) were recruited from the outpatient autism clinic at the MIND Institute (University of California, Davis).
Groups:
- Hyperbaric Oxygen Treatment (HBOT): Subjects received a total of 80 days (therefore, 80 treatments) over 20 weeks: 40 days of Hyperbaric Oxygen Treatment (HBOT) (1.5 atmosphere absolute; 100 percent oxygen) for 1 hour, 5 days a week for 8 weeks, followed by a 4 week break, and then another 40 days of HBOT over 8 weeks.
Period: First 8 Weeks (40 Treatments)
Arm/Group | Hyperbaric Oxygen Treatment (HBOT)
Started | 10
Completed | 10
Not Completed | 0
Period: 4-Week Break From Treatment
Arm/Group | Hyperbaric Oxygen Treatment (HBOT)
Started | 10
Completed | 10
Not Completed | 0
Period: Second 8 Weeks (40 Treatments)
Arm/Group | Hyperbaric Oxygen Treatment (HBOT)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyperbaric Oxygen Treatment (HBOT)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 5.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Given Clinical Global Impression Scale - Improvement (CGI-I) Score
Description: Assessment of global changes in severity of autistic symptoms. CGI-I scores formulated by the clinician based on parent interview of changes in the child's behavior and from direct clinical observation, where scores of 0 = no improvement,1 = minimally improved, 2 = much improved, and 3 = very much improved.
Time Frame: Baseline, 8 Weeks from baseline, and 20 Weeks from baseline
Measure: Number; unit: participants
Arm/Group | Hyperbaric Oxygen Treatment (HBOT)
Number analyzed (Participants) | 10
participants
  CGI-I Score of exactly 1 at 40 days | 5
  CGI-I Score of exactly 2 at 40 days | 5
  CGI-I Score of exactly 2 at 80 days | 10

ADVERSE EVENTS:
Arm/Group | Hyperbaric Oxygen Treatment (HBOT)
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen Treatment (HBOT) (N=10)
Seizure (Nervous system disorders) | 1 (1) — Likely not related to HBOt treatment. Only ear pain, increased fatigue, dehydration, and increased mouthing of objects were judged to be likely related to the HBOT treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen Treatment (HBOT) (N=10)
Ear Discomfort (Ear and labyrinth disorders) | 3 (3)
Ear Infection (Ear and labyrinth disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
1) Small sample size 2) Lack of control group prevented an examination of whether changes in clinical measure of disease severity were due to HBOT or other factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No